CLINICAL TRIAL: NCT07349563
Title: Effect of Nature-Based Virtual Reality and Two-Dimensional Nature Videos on OSCE-Related Exam Stress in Nursing Students: A Randomized Controlled Trial
Brief Title: Effects of Nature-Based Virtual Reality and 2D Nature Videos on OSCE Exam Stress in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Güzin Ünlü Suvari, Lecturer, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-15/572
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stress; Virtual Reality; Students; Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-Based Virtual Reality (Experimental): Participants receive a brief nature-based virtual reality relaxation session prior to the OSCE examination.
  Interventions: Other: Nature-Based Virtual Reality
- 2D Nature Video (Experimental): Participants watch a two-dimensional nature video for relaxation prior to the OSCE examination.
  Interventions: Other: 2D Nature Video

INTERVENTIONS:
Other: Nature-Based Virtual Reality — Participants in the intervention group will receive a short nature-based virtual reality relaxation session prior to the OSCE examination. The VR content consists of calming natural environments with gentle visual transitions and ambient sounds designed to promote relaxation and reduce stress. The session is delivered using a head-mounted display and lasts approximately 5-10 minutes.
  Arms: Nature-Based Virtual Reality
Other: 2D Nature Video — Participants in the control group will watch a two-dimensional nature video prior to the OSCE examination. The video presents relaxing natural scenes accompanied by ambient sounds and is displayed on a standard screen for approximately 5-10 minutes as a non-immersive relaxation intervention.
  Arms: 2D Nature Video

SUMMARY:
Objective Structured Clinical Examinations (OSCEs) are widely used in nursing education to assess clinical skills but are known to induce significant psychological and physiological stress due to performance anxiety, time pressure, and observation. Exam-related stress has been associated with changes in heart rate variability (HRV), particularly increased low-frequency/high-frequency (LF/HF) ratios, reflecting heightened sympathetic activity. Such stress may negatively affect cognitive performance, clinical competence, and professional readiness.

Nature-based virtual reality (VR) has emerged as a promising intervention for stress reduction by providing immersive, calming environments that promote relaxation and autonomic regulation. Previous studies suggest that short VR-based nature sessions can effectively reduce anxiety and may be more effective than two-dimensional (2D) nature videos, which represent a more accessible but less immersive alternative. However, evidence regarding the use of VR and 2D nature videos for managing stress during high-stakes clinical examinations such as OSCEs is limited.

This randomized controlled study aims to compare the effectiveness of nature-based VR and 2D nature videos in reducing OSCE-related stress among third-year nursing students using physiological (PPG-derived LF/HF ratio) and subjective (STAI and SUD) outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate third-year nursing students scheduled to take the final OSCE examination.
* Aged between 18 and 25 years.
* Considered healthy, with no known cardiovascular disease or chronic stress-related disorders.
* Willing to participate in the virtual reality or 2D nature video intervention.
* Able to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Known sensitivity or intolerance to virtual reality, including symptoms such as dizziness, nausea, headache, or visual discomfort.
* Medical conditions that may affect photoplethysmography (PPG) measurements, such as cardiac arrhythmias or significant skin sensitivity at the measurement site.
* Use of medications that may influence heart rate variability, including beta-blockers.
* Inability to allocate sufficient time to participate in the pre-examination stress management intervention.
* Pregnancy, acute illness, or current use of psychiatric medications.
* Refusal to participate or failure to provide informed consent.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
State Anxiety (STAI-State Score) | Baseline (pre-intervention, before OSCE) and immediately after the OSCE examination (post-OSCE).
  Change in state anxiety levels measured using the State-Trait Anxiety Inventory (STAI-State) to evaluate OSCE-related anxiety in nursing students.
Subjective Distress (SUD Score) | Baseline (pre-intervention), immediately after the intervention (post-intervention), and immediately after the OSCE examination (post-OSCE).
  Change in subjective stress levels assessed using the Subjective Units of Distress Scale (SUD).
Physiological Stress Response (LF/HF Ratio) | Baseline (pre-intervention) and immediately after the intervention (post-intervention).
  Change in physiological stress response assessed by heart rate variability (HRV), expressed as the low-frequency/high-frequency (LF/HF) ratio derived from photoplethysmography (PPG) recordings.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared due to privacy concerns and the sensitive nature of maternal and infant health information. However, anonymized data may be made available upon reasonable request to the corresponding author after publication of the study results.

REFERENCES:
- [Background] Camara, D., & Hicks, R. E. (2019). Using virtual reality to reduce state anxiety and stress in University students: An experiment. Global Science and Technology Forum (GSTF) Journal of Psychology, 4(1).
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Namvari M, Lipoth J, Knight S, Jamali AA, Hedayati M, Spiteri RJ, Syed-Abdul S. Photoplethysmography Enabled Wearable Devices and Stress Detection: A Scoping Review. J Pers Med. 2022 Oct 31;12(11):1792. doi: 10.3390/jpm12111792. PMID 36579537
- [Background] Liu, K. Y., Ponnapalli, P., & Dwivedi, A. K. (2025). Design of a Low-Cost Wearable System for Long-Term Continuous Heart Rate Monitoring. In Advances in Intelligent Systems (pp. 299-311). Apple Academic Press.
- [Background] Puleo, S., Diana, G., Pasta, S., Scardulla, F., & D'Acquisto, L. (2024, September). Sensor-based bioprosthetic valve monitoring: Numerical simulation and experimental design. In International Conference of the Italian Association of Design Methods and Tools for Industrial Engineering (pp. 44-51). Cham: Springer Nature Switzerland.
- [Background] Lundin RM, Yeap Y, Menkes DB. Adverse Effects of Virtual and Augmented Reality Interventions in Psychiatry: Systematic Review. JMIR Ment Health. 2023 May 5;10:e43240. doi: 10.2196/43240. PMID 37145841
- [Background] Riches S, Azevedo L, Bird L, Pisani S, Valmaggia L. Virtual reality relaxation for the general population: a systematic review. Soc Psychiatry Psychiatr Epidemiol. 2021 Oct;56(10):1707-1727. doi: 10.1007/s00127-021-02110-z. Epub 2021 Jun 13. PMID 34120220
- [Background] Mazgelyte E, Rekiene V, Dereskeviciute E, Petrenas T, Songailiene J, Utkus A, Chomentauskas G, Karciauskaite D. Effects of Virtual Reality-Based Relaxation Techniques on Psychological, Physiological, and Biochemical Stress Indicators. Healthcare (Basel). 2021 Dec 14;9(12):1729. doi: 10.3390/healthcare9121729. PMID 34946455
- [Background] Nafee, H. M., Ahmed, A. E. S., & Hussien, A. M. (2019). Objective structured clinical examination versus traditional clinical examination among nursing students: A comparative approach. Journal of Nursing Education and Practice, 9(2), 42-52.
- [Background] Ratanasiripong P, Park JF, Ratanasiripong N, Kathalae D. Stress and Anxiety Management in Nursing Students: Biofeedback and Mindfulness Meditation. J Nurs Educ. 2015 Sep;54(9):520-4. doi: 10.3928/01484834-20150814-07. PMID 26334339
- [Background] Xu J, Khanotia A, Juni S, Ku J, Sami H, Lin V, Walterson R, Payne E, Jo H, Rahimpoor-Marnani P. Effectiveness of Virtual Reality-Based Well-Being Interventions for Stress Reduction in Young Adults: Systematic Review. JMIR Ment Health. 2024 Mar 29;11:e52186. doi: 10.2196/52186. PMID 38551625